CLINICAL TRIAL: NCT00166699
Title: The Clinical Evaluation of a Novel Ultrasound Probe to Guide the Insertion of Central Regional Anaesthesia Using a Regional Anaesthetic Needle Modified to Aid Insertion Under Ultrasound Guidance in Morbidly Obese Women Undergoing Elective Caesarean Section
Brief Title: A Trial of the Use of Ultrasound to Aid the Insertion of Combined Spinal Epidural Anaesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: erica packard, North Glasgow University NHS Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04AN003(1); rec reference number04AN003(1)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Obesity; Pregnancy
Keywords: ultrasonography; obesity; Cesarean Section; Anesthesia; Epidural
MeSH Terms: conditions — Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation (No Intervention): Use of palpation to guide the the insertion site of combined spinal epidural needle in obese parturients
- ultrasound (Experimental): The use of ultrasound to guide the insertion of a combined spinal epidural needle
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — The use of ultrasound to guide the insertion of combined spinal epidural needle
  Other Names: Split array transducer
  Arms: ultrasound

SUMMARY:
The study will establish whether the use of ultrasound scanning with a purpose built probe will aid the insertion of the needles for epidural and spinal anaesthesia for obese women undergoing elective caesarean section The study group will be 46 obese women (defined by the ratio of height to weight) at time of initial booking ultrasound scan, undergoing routine caesarean section with no serious illnesses that are both willing and able to provide informed consent prior to spinal epidural anaesthesia. Patients will be excluded if they have signs or symptoms of systemic or local infection, if they have a history of previous spinal surgery, a blood clotting abnormities.

In order to evaluate the clinical usefulness of the ultrasound probe a randomised comparison of the traditional clinical methods of feeling the bones of the spine and ultrasound guided insertion of a combined spinal epidural anaesthetic will be undertaken. The rodiera tiped 17/18G 90mm tuohy needle and 123mm 27G spinal needle manufactured by Sarstedt will be the regional needles used for the combined spinal epidural anaesthetic. Randomisation into two groups (ultrasound guided needle insertion and feeling the bones) will be by computer generated random sequence. This information will be recorded in sealed envelopes and placed in the ward. Patients who meet the inclusion criteria and who consent immediately prior to caesarean section will be sequentially assigned a number that will correspond to a sealed envelope. The main aim of the study will be to detect any difference in time taken to insert epidural catheter via the needle in the patients back. The other factors measured will be the number of times the skin is punctured and bone touched by the needle, number of conversions from regional (spinal epidural) to general anaesthesia, patient satisfaction scores, requirement for extra local anaesthetic following initial blockade during Caesarean section.

The factors will be compared by student t-test using Statistica6 (StatSoft,Inc.(2001). STATISTICA (data analysis software system), version 6. www.statsoft.com). A population of 46 patients will be required assuming a mean time for inserting a combined spinal epidural without

DETAILED DESCRIPTION:
Study objective:

The clinical evaluation of a novel ultrasound probe to guide the insertion of central regional anaesthesia using a regional anaesthetic needle modified to aid insertion under ultrasound guidance in morbidly obese women undergoing elective caesarean section. - (full title) The clinical evaluation of a novel ultrasound probe-(short title)

Background and Rationale:

Cases of trauma to the conus medularis following spinal anaesthesia have been highlighted recently by Reynolds1. A second report in the same vein described the inaccuracy of using Tuffier's line between the iliac crests to identify a safe lumbar interspace2. As suspected by many clinicians, precise lumbar interspace identification by palpation is prone to error. Broadbent2 et al confirmed this showing that anaesthetists were only 29% accurate, as determined by MRI/ (Ultrasonography was not investigated by Broadbent). The inaccuracy was corroborated by Furness et al3. who showed that clinical identification by anaesthetists using palpation was 30% accurate, as assessed by lumbar spine X-ray. In contrast, in the latter study, placement of markers using ultrasonography at L3-4 interspace was 71% accurate, a figure which is comparable with the 76% accuracy in the preliminary study described below . It should be noted in the Furness study that ultrasonography was performed by a consultant radiologist but in our study an anaesthetist performed the procedure. The Broadbent and Furness studies both documented that identification by anaesthetists using palpation was often inaccurate by two, three or four interspaces. Using ultrasound, in both the Furness3 study and our study, markers were always within one interspace of the intended position.

Morbid obesity is an increasingly prevalent problem in obstetric practice. Landmarks are often impalpable in obese patients making insertion of epidurals problematic. Thus there is clear clinical need to develop a safe efficient way to administer epidural anaesthesia. The central hypothesis of our application is that ultrasonic visualisation of the landmarks will aid insertion. Further it is possible to develop and manufacture a probe for general use by anaesthetists that will improve current clinical practice in this problematic area.

Initial study to investigate accuracy ultrasound by non radiologist:

An exploratory study was undertaken to determine the precision with which an anaesthetist could identify the correct L3-4 interspace using ultrasonography. Twenty-three ultrasonographic examinations of lumbar spine were performed by an anaesthetic senior house officer with minimal training on patients undergoing an elective MRI scan of the lumbar spine. Seventeen patients were eligible for inclusion in this study. Patients' median age was 47 years, and body mass index 27 kg/m2. In 13 of the 17 (76%) patients, the SHO using ultrasonography was able to place a marker correctly at the L3-4 interspace as indicated by MRI. In four patients, the marker was at the L2-3 interspace. In five of the 17 patients apposition of spinous processes was noted on MRI scan and it was in three of these patients that the marker was at the L2-3 interspace.

Ultrasound has been used to aid the insertion of central neuraxial anaesthesia on three occasions. (Watson et al unpublished). The 3 cases below describe the successful ultrasound assisted insertion of three neuroaxial blocks to allow both emergency and elective caesarean section. The first two reports are based on the same woman undergoing emergency and elective section during two consecutive pregnancies complicated by obesity and pre-eclampsia. The third case report was complicated by the previous spinal fusion surgery for a lumbar disc prolapse.

Aim:

To determine if the novel ultrasound transducer provides a method of reducing the time taken to insert a combined spinal epidural anaesthetic in obese women undergoing elective caesarean section

Study population:

Sample Population:

The maternity hospitals involved in this trial have in excess of 25,000 deliveries per year and a significant percentage of these mothers come from under privileged backgrounds with a high incidence of morbid obesity. A study population of 46 patients will be recruited from those women undergoing elective caesarean section

Study procedures

Randomisation of patients:

Randomisation into two groups will be by computer generated block randomisation method. This information will be recorded in sealed envelopes and placed in the labour ward at princess royal maternity. Patients who meet the inclusion criteria and who consent will be sequentially assigned a number that will correspond to a sealed envelope.

Method:

Prior to the study starting we will recruit and consent 10 elective section patients to optimise the quality control of for imaging with the split array ultrasound transducer.

In order to evaluate the clinical efficacy of the ultrasound probe a randomised comparison of the traditional clinical methods of palpation and ultrasound guided insertion of a (CSE)combined spinal/epidural anaesthetic will be undertaken. The combined spinal epidural (17/18G 90mm rodiera tiped tuohy needle and 123mm 27G spinal needle manufactured by Sarstedt will be used for all patients and all the tuohy needles will be sand and bead blasted, desterilised and repackaged prior to use. All patients will have a spinal anaesthetic 2.4mls of heavy bupivacaine and a 22G epidural catheter sited via a 16G tuohy needle with diamorphine or fentanyl. All anaesthetic procedures will be undertaken by the same experienced anaesthetist. However those patients in the ultrasound group will have the insertion of the tuohy needle guided by ultrasound and the will be compared to the current method of palpation. All patients will then undergo elective caesarean section. Patient's having an ultrasound inserted using palpation may be transferred to the ultrasound guided group after 30 minutes of attempted insertions or at the discretion of the anaesthetist treating the patient.

Withdrawal of patients from study:

Any patient may withdraw from the study at any time without giving any reason or justification.

Any protocol violation will result in the patient being immediately withdrawn from the study If the patient requires emergency caesarean section they will be withdrawn from the study If the patient is in labour prior to their intended date of operative delivery they will be withdrawn from the study Any patient who does not undergo an caesarean section will be withdrawn from the study

Statistical considerations:

Primary end points:

The primary end point will be time taken to insert an epidural catheter.

Secondary end points:

The number of times the skin is punctured The number of times the cortex of bone touched by the epidural needle The number of conversions from regional (central-neuraxial) to general anaesthesia Patient satisfaction scores immediately post op and at 30 minutes post op The volume and concentration of supplementary local anaesthetic administration following primary spinal blockade during caesarean section Number of needle advancements

Number of conversions to general anaesthesia

Number of 'dry spinal taps'

Patient numbers:

A population of 46 patients will be required assuming a mean time for inserting a combined spinal epidural without ultrasound guidance of 15 minutes and with ultrasound guidance of 10 minutes with a standard deviation of 5 minutes for both groups ( power=90%, alpha error =0.05).

Assessment of Safety and Efficacy:

The time taken to perform the CSE will be recorded from the moment the skin is sterilised to the moment the epidural catheter has been fixed to the skin. A record of the number of attempts and number of times bone is encountered by the needle will be recorded. If patients in the palpation group require ultrasound assistance to locate the epidural space this will also be recorded. Drugs administered both systemically and intrathecally or epidurally will be documented. Patients will be assessed immediately after insertion of the CSE with regard to comfort during the procedure and and pain experienced. They shall also be reassessed 30 minutes postoperatively to ascertain their overall satisfaction of the technique for the surgery, to ensure no pain was experienced during the operation. They should also be visited on the first postoperative day, specifically to look for any complications of the CSE such as headache or neuropraxia, and should receive a final check prior to discharge at 5 days to ensure no adverse events have occurred.

ELIGIBILITY:
Inclusion Criteria:

* Elective Caesarean section > 38/52 gestation
* BMI at booking scan (circia 13/52 gestation)>=35
* ASA = 1,2 or 3 patients only

Exclusion Criteria:

* Abnormal clotting screen (coagulopathy) or thrombocytopenia ( < 100,000)
* Unable to give informed consent to combined spinal epidural anaesthesia
* Previous spinal surgery or known spinal pathology
* Signs, symptoms or laboratory evidence of local infection or systemic sepsis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary end point will be time taken to insert an epidural catheter. | During the c-section

SECONDARY OUTCOMES:
The number of times the skin is punctured | anaesthesia induction
The number of times the cortex of bone touched by the epidural needle | anaesthesia induction
The number of conversions from regional (central-neuraxial) to general anaesthesia | anaesthesia induction
Patient satisfaction scores immediately post op and at 30 minutes post op | 30mins post operatively
The volume and concentration of supplementary local anaesthetic administration following primary spinal blockade during caesarean section | intraoperatively
Number of needle advancements | Induction of anaesthesia
Number of conversions to general anaesthesia | induction of anaesthesia
Number of 'dry spinal taps' | induction of anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: malcolm J watson, MBCHB, Principal Investigator — North Glasgow University Hospitals Division
Locations (5):
- United Kingdom (5):
  - Princess Royal maternity, Glasgow, Scotland
  - Queen mother's maternity, Glasgow, Scotland
  - Southern general maternity hospital, Glasgow, Scotland
  - Paisley maternity hospital, Paisley, Scotland
  - Wishaw Maternity hospital, Wishaw, Scotland